CLINICAL TRIAL: NCT00393393
Title: A Single-Blind Prospective Parallel Control Group Pilot Study to Assess the Effect of Hylan G-F 20 (Synvisc) Supplementation on Cartilage Preservation in Osteoarthritis of the Knee
Brief Title: Effectiveness Study of Hylan G-F 20 to Preserve Cartilage in Osteoarthritis of the Knee
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cabrini Medical Centre (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 05-11-07-05
Record Dates: First submitted 2006-10-26; First posted 2006-10-27 (Estimated); Last update posted 2006-10-27 (Estimated); Status verified 2006-10

CONDITIONS: Osteoarthritis
Keywords: osteoarthritis; knee; hylan
MeSH Terms: conditions — Osteoarthritis

INTERVENTIONS:
Drug: intra-articular injection of Hylan G-F 20

SUMMARY:
That Hylan G-F 20 may act to protect cartilage from the expected degree of degradation over a 12 month period in subjects with moderate to marked osteoarthritis of the knee

DETAILED DESCRIPTION:
Two courses of Hylan G-F 20 ( Synvisc) administered by intra-articular injection at 6 monthly intervals. MRI examinations of the knee for estimation of cartilage volume prior to treatment, before second course and at 12 months in 40 subjects with Grade 2/3 osteoarthritis of knee . A further 40 subjects with similar degree of osteoarthritis of knee who do not receive Hylan G-F therapy will be assessed by MRI in identical manner.

ELIGIBILITY:
Inclusion Criteria:

* grade 2 or 3 osteoarthritis knee age 18 - 80 pain score VAS >39 mm on 100mm scale

Exclusion Criteria:

* surgery in prior 12 months significant valgus deformity recent trauma use of opioid analgesia unstable medical condition recent corticosteroid injection morbid obesity

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2006-01; Study Completion 2006-01

PRIMARY OUTCOMES:
Cartilage volume as assessed by magnetic resonance imaging

CONTACTS AND LOCATIONS:
Overall Officials: stephen hall, MBBS, FRACP, Principal Investigator — Cabrini Medical Centre
Locations (1):
- Emeritus Research, Malvern, Victoria, Australia

REFERENCES:
- [Derived] Wang Y, Hall S, Hanna F, Wluka AE, Grant G, Marks P, Feletar M, Cicuttini FM. Effects of Hylan G-F 20 supplementation on cartilage preservation detected by magnetic resonance imaging in osteoarthritis of the knee: a two-year single-blind clinical trial. BMC Musculoskelet Disord. 2011 Aug 24;12:195. doi: 10.1186/1471-2474-12-195. PMID 21861935